CLINICAL TRIAL: NCT03155204
Title: Phase I Randomised, Five-period Cross-over Study in Healthy Male and Female Volunteers to Compare the Pharmacokinetics of Tiotropium Delivered From Four Test pMDI Products With Spiriva Respimat
Brief Title: Comparison of the Pharmacokinetics of Tiotropium Delivered From Test Inhaler Products With A Reference Product
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CSP-07-000039
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: inhalation; LABA; corticosteroid
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Test Product 1 (Experimental): tiotropium pMDI 2 inhalations
  Interventions: Drug: tiotropium pMDI
- Test Product 2 (Experimental): tiotropium pMDI 2 inhalations
  Interventions: Drug: tiotropium pMDI
- Test Product 3 (Experimental): tiotropium pMDI 2 inhalations
  Interventions: Drug: tiotropium pMDI
- Test Product 4 (Experimental): tiotropium pMDI 2 inhalations
  Interventions: Drug: tiotropium pMDI
- Commercial Product (Active Comparator): tiotropium Respimat 2 inhalations
  Interventions: Drug: tiotropium pMDI

INTERVENTIONS:
Drug: tiotropium pMDI — inhalation
  Other Names: Spiriva Respimat

SUMMARY:
The purpose of this study is to compare the absorption of four different inhalation products with the reference product in healthy volunteers.

DETAILED DESCRIPTION:
Healthy subjects will be enrolled and will receive single doses of 4 test inhalation products and one reference inhalation product according to a five-period cross-over design. Plasma tiotropium levels will be measured pre-dose and over 8 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer
* Willing and able to give informed consent
* Willing to withhold all alcoholic beverages for 48 hours and all xanthine- containing foods and beverages for 24 hours prior to reporting to clinic
* Subjects must agree to use an adequate method of contraception from admission through 12 weeks after last administration

Exclusion Criteria:

* Evidence or history of clinically significant abnormalities or disease or chronic respiratory disorders
* Any presence or history of a clinically significant allergy including any adverse reaction to study drug
* History of drug or alcohol abuse within the past 2 years
* Smoked tobacco within the past 6 months or have a history of more than 10- pack years (number of packs smoked per day x number of years smoked)
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Have received any prescription medication within 4 weeks or investigational medication within 12 weeks of study (exception: contraceptives are permitted)
* Have received any non-prescription medication within 14 days prior to dosing (exception: paracetamol use within 2 days)
* Upper respiratory tract infection (excluding otitis media) within 14 days of the first study day, or lower respiratory tract infection within the last 3 months
* If female, nursing, lactating or pregnant
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 24 hr
  noncompartmental analysis

SECONDARY OUTCOMES:
Adverse events | 24 hr
  reported adverse events
Area Under the Plasma Concentration vs Time Curve (AUC) | 24 hr
  trapezoidal rule

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Sessions, PhD, Study Chair — 3M
Locations (1):
- 3M Health Care, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No
publication